CLINICAL TRIAL: NCT03186378
Title: A Phase 2, Open-Label Study to Evaluate the Safety, Efficacy and Systemic Exposure of VP-102 Topical Film Forming Solution [0.7% (w/v) Cantharidin] in Subjects (2 Years and Older) With Molluscum Contagiosum
Brief Title: Evaluation of Systemic Exposure to VP-102 in Subjects With Molluscum Contagiosum.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Verrica Pharmaceuticals Inc. (Industry)
Collaborators: Paidion Research, Inc. (Industry); Database Integrations, Inc. (Industry); Cato Research (Industry); Instat Services (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VP-102-103
Record Dates: First submitted 2017-06-12; First posted 2017-06-14 (Actual); Results first posted 2021-08-09 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-08

CONDITIONS: Molluscum Contagiosum
MeSH Terms: conditions — Molluscum Contagiosum | interventions — VP-102

STUDY DESIGN:
Intervention Model Description: Open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Exposure Group (Experimental): This group is open label and allows for up to 16 subjects with 21 or more molluscum lesions will be enrolled. They must complete all blood draws or will be replaced. Intervention Drug: Subjects will receive treatment to their molluscum contagiosum lesions per protocol with VP-102 using the VP-102 applicator.
  Interventions: Combination Product: VP-102 with applicator
- Standard Group (Experimental): This group is open label allowing up to 16 subjects with 20 lesions or less to be enrolled. Drug: Subjects will receive treatment to their molluscum lesions with VP-102 using the VP-102 applicator.
  Interventions: Combination Product: VP-102 with applicator

INTERVENTIONS:
Combination Product: VP-102 with applicator — Subjects will receive treatment to their molluscum contagiosum with VP-102.

SUMMARY:
The primary objective of the study is to determine the presence or absence of systemic cantharidin exposure from a single 24-hour dermal application of VP-102 topical film-forming solution [0.7% (w/v) cantharidin] (VP-102) when applied to molluscum contagiosum (molluscum) lesions on pediatric subjects 2 years old and older. Treatment will continue over the course of 3 additional 21 day intervals allowing for further evaluation of safety, efficacy and impact on quality of life.

DETAILED DESCRIPTION:
This is a Phase 2, Open-Label Study to Evaluate the Safety, Efficacy and Systemic Exposure of VP-102 Topical Film Forming Solution [0.7% (w/v) cantharidin] in subjects 2 years and older with Molluscum Contagiosum. Up to 40 subjects will be enrolled in the study with the goal of 16 meeting criteria for, and completing all scheduled blood draws outlined in the exposure portion of the trial. Subjects that do not have enough molluscum lesions to participate in the exposure study but do meet all other criteria to participate in the study will be enrolled in the standard treatment group. No more than 16 subjects will complete exposure group activities; up to 16 subjects will be enrolled in the standard treatment group. The additional 8 subjects may be used for replacement patients. At least 3 patients in the exposure group will be from 2-5 years of age. All subjects will receive VP-102 containing 0.7% cantharidin to molluscum lesions every 21 days for a maximum of 4 sessions or until complete clearance.

In the exposure group, blood samples for systemic exposure evaluation will be collected on Day 1, prior to the drug application, and 2 (± 30 minutes), 6 (± 1 hour) and 24 (±3 hours) hours post-application. A dermatological examination will be performed by a qualified investigator quantifying molluscum lesion counts at every study visit.

ELIGIBILITY:
Inclusion Criteria:

1. Be healthy subjects ages 2 years and older.
2. Patients with 1-20 lesions may be enrolled and treated in the standard treatment group but are not eligible for the exposure study.
3. Patients with 21 or more lesions may only be enrolled in the exposure group. Subjects participating in the Exposure group must have at least 21 lesions treated at Day 1 to qualify.
4. Be otherwise medically healthy with no clinically significant medical history as determined by the investigator. Patients exhibiting active Atopic Dermatitis may be enrolled.
5. Refrain from application of all topical agents including alcohol-based sanitary products and sunscreens for a minimum of 4 hours before Study drug application. Topical agents including alcohol-based sanitary products and sunscreens may be used after application of the study drug so long as they are not applied to or near treated skin.
6. Refrain from swimming, bathing or prolonged immersion in water until the Study drug is removed.
7. Have the ability or have a guardian able to follow study instructions and be likely to complete all study requirements.
8. Provide assent in a manner approved by the institutional review board (IRB) and have a parent/guardian provide written informed consent as evidenced by signature on IRB approved assent/consent forms.
9. Provide written authorization for use and disclosure of protected health information.
10. Agree to allow photographs of all selected lesions to be taken and/or send photos via text or email to the study team for assessment at 24 hours post treatment. Photos may be used as part of the study data and/or marketing package. (Photographs will be de-identified to those outside the research team. Effort will be made to ensure that no photos with identifiable features are obtained).

Exclusion Criteria:

1. Are unable to cooperate with the requirements or visits of the study, as determined by the investigator.
2. Have molluscum venereum (sexually transmitted molluscum).
3. Have active molluscum eczema.
4. Are systemically immunosuppressed or are receiving treatments such as chemotherapy or other non-topical immunosuppressive agents.
5. Have had any previous treatment of molluscum in the past 14 days including the use of cantharidin, antivirals, retinoids, curettage or freezing of lesions. Additional treatments for molluscum should not be implemented during the course of the study.
6. Have history of illness or any dermatologic disorder, which, in the opinion of the investigator will interfere with accurate counting of lesions or increase the risk of adverse events.
7. History or presence of clinically significant medical, psychiatric, or emotional condition or abnormality that in the opinion of the investigator would compromise the safety of the subject or the quality of the data.
8. Have a history or presence of hypersensitivity or an idiosyncratic reaction to the Study drug or related compounds, or drug product excipients.
9. Have a condition or situation that may interfere significantly with the subject's participation in the study (e.g., patients who required hospitalization in the 2 months prior to screening for an acute or chronic condition including alcohol or drug abuse), at the discretion of the investigator.
10. Have received another investigational product within 14 days prior to the first application of the Study drug.
11. Have been treated within 14 days with a product that contains the active ingredient in VP-102 (topical or homeopathic preparations) for any reason prior to screening.
12. Are sexually active or may become sexually active and are unwilling to practice responsible birth control methods. Females that have reached menarche, must have a negative urine pregnancy test at screening and each visit prior to treatment with study medication.
13. Are pregnant or breastfeeding.

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-06-08 (Actual); Primary Completion 2018-06-25 (Actual); Study Completion 2018-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Goldenberg, MD, Study Director — Verrica Pharmaceuticals Inc.
Locations (1):
- Midwest Children's Health, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Niazi S, Brabec B, Anschutz L, Willson C, Davidson M, Burnett P. A Phase 2 Open-Label Study to Evaluate VP-102 for the Treatment of Molluscum Contagiosum. J Drugs Dermatol. 2021 Jan 1;20(1):70-75. doi: 10.36849/JDD.5626. PMID 33400412

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Exposure Group | Standard Group
Started | 17 | 16
Completed | 16 | 16
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: ITT Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Exposure Group | Standard Group | Total
Number analyzed (Participants) | 17 | 16 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.6 (3.45) | 6.8 (3.15) | 6.7 (3.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 10 | 8 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 17 | 14 | 31
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 16 | 14 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17 | 16 | 33
Baseline Number of Molluscum Lesions [Mean (Standard Deviation); unit: molluscum lesions] | 47.4 (25.69) | 11.6 (6.33) | 30.0 (26.07)

OUTCOME MEASURES:

1. Primary Outcome: The Presence or Absence of Systemic Exposure to Cantharidin by the Collection and Analysis of Plasma Samples From Patients With 21 or More Molluscum Lesions Following Treatment of VP-102.
Description: The primary objective is to determine any potential systemic exposure from a single 24-hour dermal application of VP-102 topical film-forming solution when applied to molluscum contagiosum (molluscum) lesions on pediatric subjects 2 years old and older.
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Exposure Group
Number analyzed (Participants) | 16
Participants
  Any Concentration Level of VP-102 above LLOQ (2.5ng/ml) Pre-treatment: Yes | 0
  Any Concentration Level of VP-102 above LLOQ (2.5ng/ml) Pre-treatment: No | 16
  Any Concentration Level of VP-102 above LLOQ (2.5ng/ml) 2hr Post Treatment: Yes | 1
  Any Concentration Level of VP-102 above LLOQ (2.5ng/ml) 2hr Post Treatment: No | 15
  Any Concentration Level of VP-102 above LLOQ (2.5ng/ml) 6hr Post Treatment: Yes | 0
  Any Concentration Level of VP-102 above LLOQ (2.5ng/ml) 6hr Post Treatment: No | 16
  Any Concentration Level of VP-102 above LLOQ (2.5ng/ml) 24hr Post Treatment: Yes | 0
  Any Concentration Level of VP-102 above LLOQ (2.5ng/ml) 24hr Post Treatment: No | 16

2. Secondary Outcome: Measurement of Efficacy - Complete Clearance
Description: Proportion of subjects exhibiting complete clearance of all treated molluscum lesions (baseline and new) on or before Week 12 (EOS).
Time Frame: Baseline through EOS Day 84
Population: Complete Clearance of Molluscum Lesions - Completer Population
Measure: Count of Participants; unit: Participants
Arm/Group | Exposure Group | Standard Group
Number analyzed (Participants) | 16 | 16
Participants
  Complete Clearance Day 21 | 0 | 3
  Complete Clearance Day 42 | 2 | 7
  Complete Clearance Day 63 | 4 | 9
  Complete Clearance EOS Day 84 | 6 | 10

3. Other Pre Specified Outcome: Proportion of Subjects Exhibiting a 90% or Greater Reduction of All Treated Molluscum Lesions (Baseline and New) at the EOS Visit.
Description: Summaries of >=90% clearance by visit include clearance at that visit or any earlier visit (cumulative) baseline and ew at the EOS visit.
Time Frame: Baseline to EOS Day 84
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Exposure Group | Standard Group
Number analyzed (Participants) | 17 | 16
Participants
  >=90% Clearance Day 21 | 0 | 3
  >=90% Clearance Day 42 | 5 | 7
  >=90% Clearance Day 63 | 8 | 10
  >=90% Clearance Day 84 | 12 | 13

4. Other Pre Specified Outcome: Percent Reduction of Treated Molluscum Lesions From Baseline at the EOS Visit.
Description: Percent reduction of treated molluscum lesions from Baseline Visit at the EOS visit.
Time Frame: Baseline to EOS Day 84
Population: ITT Population
Measure: Mean (Standard Deviation); unit: percentage change from Baseline
Arm/Group | Exposure Group | Standard Group
Number analyzed (Participants) | 16 | 16
percentage change from Baseline | -87.8 (21.25) | -93.0 (12.93)

5. Other Pre Specified Outcome: Change From Baseline in the Number of Treated Molluscum Lesions at the EOS Visit.
Description: Molluscum Lesions- Change from Baseline visit in the number of treated molluscum lesions at the EOS Day 84 visit
Time Frame: Baseline to EOS Day 84
Population: ITT Population
Measure: Mean (Standard Deviation); unit: change in wart count
Arm/Group | Exposure Group | Standard Group
Number analyzed (Participants) | 16 | 16
change in wart count | -39.3 (21.98) | -10.7 (6.16)

6. Other Pre Specified Outcome: Change From Baseline in Quality of Life and Impact of Skin Disease as Measured by CDLQI Assessment
Description: Change from Baseline in quality of life and impact of skin disease as measured by CDLQI assessment, Children's Dermatology Life Quality Index (CDLQI)- Composite Score
  The CDLQI was a 10-item questionnaire completed by subject/parent to assess skin condition over the previous week. From responses to that questionnaire, a composite score was calculated. The calculated composite score was the sum of the individual 10 items of the CDLQI and could range from 0-30. For each item on the CDLQI, a score of 0-3 was assigned using the following scores per response:
  * 3: Very much (or Prevented School, Question 7 only)
  * 2: Quite a lot
  * 1: Only a little
  * 0: Not at all
Time Frame: Baseline to EOS Day 84
Population: ITT Population
Measure: Mean (Standard Deviation); unit: units on a scale change from Baseline
Arm/Group | Exposure Group | Standard Group
Number analyzed (Participants) | 17 | 16
units on a scale change from Baseline | 2.71 (2.801) | 2.44 (4.115)

7. Other Pre Specified Outcome: Spread to Siblings as Measured by Any New Occurrence of Molluscum in Siblings of the Subject.
Description: Spread of molluscum to siblings as measured by any new occurrence of molluscum in siblings of the subject.
Time Frame: Baseline to EOS Day 84
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Exposure Group | Standard Group
Number analyzed (Participants) | 17 | 16
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline to EOS Day 84
Description: Adverse events summaries will only consider (TEAEs). TEAEs are defined as those AEs that occurred after dosing and those existing AEs that worsened during the study. If it cannot be determined whether the AE is treatment emergent due to an incomplete onset date, the AE will be considered to be treatment emergent.
Arm/Group | Exposure Group | Standard Group
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/16
Other Adverse Events (participants affected / at risk) | 16/17 | 13/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Exposure Group (N=17) | Standard Group (N=16)
Pain (General disorders) | 11 | 8 — General disorders and administration site conditions
Burning Sensation (General disorders) | 1 | 0 — General disorders and administration site conditions
Pyrexia (General disorders) | 1 | 0 — General disorders and administration site conditions
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Influenza (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Scar (Skin and subcutaneous tissue disorders) | 3 | 1
Application site vesicles (Skin and subcutaneous tissue disorders) | 1 | 0
Cellulitis (Skin and subcutaneous tissue disorders) | 1 | 0
Impetigo (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Subcutaneous abscess (Skin and subcutaneous tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 3
Vomiting (Gastrointestinal disorders) | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Tinea infection (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Adjustment disorder (Psychiatric disorders) | 1 | 0
Lethargy (Psychiatric disorders) | 1 | 0
Tic (Psychiatric disorders) | 1 | 0
Asthma (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Administration site pain (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Eye infection (Eye disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI is bound to terms and conditions of a Sponsored Clinical Trial Agreement which has strict confidentiality obligations running to Sponsor and broad provisions restricting PI's rights to publish or present any data or Study Results without Sponsor's express review consent and review.

DOCUMENTS (2):
  • Study Protocol (2017-08-08): https://cdn.clinicaltrials.gov/large-docs/78/NCT03186378/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-04): https://cdn.clinicaltrials.gov/large-docs/78/NCT03186378/SAP_001.pdf